Abdominal hysterectomy and bilateral Magnesium sulfate infusion in oophorectomy surgery perioperative Study on "opioid consumption and its effect on postoperative analgesia

The primary outcome of this study was total iv fentanyl consumption in the first 24 hours after surgery . For an effective analgesia method, a decrease of at least 20% in 24-hour opioid use is required (1). In the independent groups t-test model created using the data of a previous similar study (2), the calculation was made by considering at least a 20% decrease in 24-hour fentanyl consumption compared to the control group as significant. In the calculation made using Cohen's D effect size of 1.318, it was calculated that 16 patients in each group should participate in the study for 95% power and maximum 5% type 1 error. Considering the possibility of dropout rate , the required sample size was calculated as 20 patients for both groups (40 patients in total).